CLINICAL TRIAL: NCT06899373
Title: Glucose Levels as a Biomaterial for Stress in Firefighters
Brief Title: Glucose Levels as a Biomarker for Stress in Firefighters
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Other Study IDs: 00182726
Record Dates: First submitted 2025-01-28; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2024-12

CONDITIONS: Stress; Sympathetic Nervous System; Hypothalamic Pituitary Adrenal
Keywords: Occupational stress; firefighter; firefighter health
MeSH Terms: conditions — Occupational Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Firefighters: 17 professional firefighters being monitored on their work shifts and days off
  Interventions: Device: Continuous glucometer

INTERVENTIONS:
Device: Continuous glucometer — The continuous glucometer is a wearable device that measures interstitial glucose levels 24 hours per day and transmits readings every one minute.

SUMMARY:
Stress is known to cause physical structures in the brain to dysregulate, resulting in health problems like cancer, cardiac disease, metabolic disorders (obesity), and depression. Firefighters experience many of these diseases at higher rates than other occupations while also experiencing highly unique stress loads. When the body's nervous system responds to stress, blood glucose levels increase. This study will equip firefighters with continuous glucometers to observe glucose levels during emergency response and other stressful events. The immediate goal of this study is to determine whether the physiological stress response of on-shift firefighters can be quantified with glucose monitoring. The long-term goal is to identify occupational firefighter stress as a health risk exposure.

DETAILED DESCRIPTION:
High morbidity conditions like suicide, cardiovascular disease, and diabetes occur at higher rates for firefighters than in other professions. Despite decades of awareness and targeted efforts to address these problems, firefighters continue to suffer from these conditions at high rates. Stress is a known contributor to these diseases in all populations, and firefighters are exposed to extremely high levels of occupational stress over a 20-30-year career. This problem is commonly approached by focusing research and interventions on the conditions themselves, but an important root cause remains understudied: activation of the sympathetic nervous system (SNS) during emergency response. This activation occurs frequently throughout a firefighter's shift and can be studied by using blood glucose levels as a surrogate marker for SNS activation. The information obtained would offer a significant perspective shift to research and intervention efforts that support firefighter health by shedding new light on SNS activation as a co-morbidity for these conditions. It would also support firefighters in managing their health by providing a new way to quantify stress exposure.

During SNS activation, the liver releases glycogen to increase blood glucose levels, fueling muscles and organs needed in a fight-or-flight response. This response is activated when firefighters are called to emergency scenes by the station alarm. The investigators will equip firefighters with continuous glucose monitors during their shifts and measure changes in serum glucose levels every minute. The hypothesis is that SNS activation will occur during emergency dispatch, resulting in increased blood glucose levels. A secondary hypothesis is that the magnitude of the glucose response will vary based on the self-reported emotional response to the call. Observing the relationship between glucose levels and SNS activation will provide a new perspective on the underlying causes of firefighter health conditions.

Aim 1: Test the hypothesis that glucose levels will increase after emergency dispatch.

Continuous glucose data will be collected every minute, allowing for the comparison of glucose levels before and after a station alarm. If the SNS is activated by a station alarm, an increase in blood glucose levels is anticipated. This information would provide insights into the frequency and magnitude of SNS activation during emergency response. This hypothesis will also generate data on variables that will be used to develop hypotheses for a subsequent study with a larger population. These variables include sleep, diet, and perceived stress. SNS activation is known to have negative health effects that contribute to chronic health problems, for which firefighters are already at elevated risk. Observing the frequency and magnitude of this nervous system response will identify an important contributor to chronic health risks for firefighters.

Aim 2: Test the hypothesis that perceived stress affects glucose levels during emergency dispatch.

Being dispatched to an emergency incident evokes an emotional and stress response that varies for each responder. The limbic system regulates emotional and stress responses, and dysregulation of this system is known to contribute to behavioral conditions. Study participants will report their perceived stress levels for each call they respond to, allowing for a comparison between perceived stress and the magnitude of glucose changes. Participants will identify the three most stressful calls during their shift and the three most stressful events during their days off. These self-reported stressful events will be used as comparison points between on-shift and off-shift stress responses. Observing the relationship between SNS activation and perceived emotional stress exposure will provide a new perspective on emotional stress experiences and help firefighters identify periods of heightened need for supportive resources.

This pilot study will generate data to inform hypotheses for a future large-scale study that may provide new directions for studying and treating chronic health conditions in firefighters. Firefighters are exposed to multiple risk factors while responding to emergency calls, increasing their likelihood of developing chronic health conditions. This study will highlight a new risk factor, enabling fire administrations, governing agencies, and firefighters to take appropriate mitigation measures. Recognizing SNS activation as a co-morbidity would support the development of new, potentially life-saving interventions and foster a cultural shift in how firefighters manage their physical and behavioral health.

ELIGIBILITY:
Inclusion Criteria:

* Full time Unified Fire Authority (UFA) employee working for a fire crew that has been designated by the UFA board as approved for study participation

Exclusion Criteria:

* Use of insulin
* Diagnosed with Diabetes Mellitus
* Practicing a ketoacidosis or intermittent fasting diet
* Intermittent use of glucocorticoids, antibiotics or benzodiazepines

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Full time firefighters that work 48 hour work shifts followed by 96 hours of rest.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in Blood Glucose Levels Following Emergency Dispatch | 2 Weeks
  Blood glucose levels will be continuously monitored every minute using continuous glucose monitors (CGMs). Glucose levels immediately before and after emergency dispatch calls will be compared to changes indicative of sympathetic nervous system (SNS) activation. The magnitude and frequency of glucose level increases will be analyzed to determine the physiological response to emergency dispatch events.
Association Between Perceived Stress and Blood Glucose Response to Emergency Dispatch | 2 Weeks
  Firefighters will self-report perceived stress levels for emergency dispatch calls. The three most stressful calls during their shift and the three most stressful events during their off-shift periods will be identified. The relationship between perceived stress ratings and changes in blood glucose levels following emergency dispatch will be analyzed to assess the impact of emotional stress on sympathetic nervous system (SNS) activation.

OTHER OUTCOMES:
Demographic and Within-Group Comparison of Blood Glucose and Perceived Stress Responses | Baseline
  Demographic variables, including age, years of service, and baseline health metrics, will be collected to assess their relationship with blood glucose responses and perceived stress levels. Within-group comparisons will be conducted to explore variations in sympathetic nervous system (SNS) activation based on individual characteristics and occupational factors.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Thiese, PhD, Principal Investigator — matt.thiese@hsc.utah.edu
Locations (1):
- Unified Fire Authority, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No
Pending participant verification